CLINICAL TRIAL: NCT05793684
Title: Phase 2 Randomized Double-Blind Placebo-Controlled Multiple-Dose 3-Period Crossover Study to Compare a Fixed Dose Combination of AD816 to Viloxazine Alone and to Placebo in Obstructive Sleep Apnea
Brief Title: AD816 Crossover Study
Acronym: VicTor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apnimed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: APV-001
Record Dates: First submitted 2023-03-18; First posted 2023-03-31 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: OSA; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Order: Period A, Period B, Period C (Experimental): The sequence of periods for each participant are assigned in random order. Each of the three crossover periods is 14 days of uninterrupted nightly dosing, with an initial lower-dose week of investigational product (IP) followed by a higher dose week (or placebo each week).
  Interventions: Drug: Period A; Drug: Period B; Drug: Period C
- Order: Period B, Period C, Period A (Experimental): The sequence of periods for each participant are assigned in random order. Each of the three crossover periods is 14 days of uninterrupted nightly dosing, with an initial lower-dose week of investigational product (IP) followed by a higher dose week (or placebo each week).
  Interventions: Drug: Period A; Drug: Period B; Drug: Period C
- Order: Period C, Period A, Period B (Experimental): The sequence of periods for each participant are assigned in random order. Each of the three crossover periods is 14 days of uninterrupted nightly dosing, with an initial lower-dose week of investigational product (IP) followed by a higher dose week (or placebo each week).
  Interventions: Drug: Period A; Drug: Period B; Drug: Period C
- Order: Period A, Period C, Period B (Experimental): The sequence of periods for each participant are assigned in random order. Each of the three crossover periods is 14 days of uninterrupted nightly dosing, with an initial lower-dose week of investigational product (IP) followed by a higher dose week (or placebo each week).
  Interventions: Drug: Period A; Drug: Period B; Drug: Period C
- Order: Period B, Period A, Period C (Experimental): The sequence of periods for each participant are assigned in random order. Each of the three crossover periods is 14 days of uninterrupted nightly dosing, with an initial lower-dose week of investigational product (IP) followed by a higher dose week (or placebo each week).
  Interventions: Drug: Period A; Drug: Period B; Drug: Period C
- Order: Period C, Period B, Period A (Experimental): The sequence of periods for each participant are assigned in random order. Each of the three crossover periods is 14 days of uninterrupted nightly dosing, with an initial lower-dose week of investigational product (IP) followed by a higher dose week (or placebo each week).
  Interventions: Drug: Period A; Drug: Period B; Drug: Period C

INTERVENTIONS:
Drug: Period A — Week 1: Viloxazine low dose + placebo; Week 2: Viloxazine high dose + placebo
Drug: Period B — Week 1: AD816 low dose; Week 2: AD816 high dose
Drug: Period C — Week 1: Placebo + Placebo; Week 2: Placebo + Placebo

SUMMARY:
The VicTor Study is a randomized, double blind, placebo-controlled, 3-period, multiple-dose crossover study in participants with OSA.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 to 75 years of age, inclusive, at the Screening Visit
2. PSG criteria (V2 only)

   1. AHI4 (Hypopneas defined by 4% oxygen desaturation) of 10-45, inclusive
   2. ≤25% of events are central or mixed apneas
3. PROMIS Fatigue or sleep related impairment or sleep disturbance (raw score): >11, i.e. at least "very mild symptoms" at V1
4. BMI between 18.5 and 40 kg/m2, inclusive

   Male participants:
5. If sexually active with female partner(s) of childbearing potential, participant must agree, from Study Day 1 through 1 week after the last dose of study drug, to practice the protocol specified contraception

   Female participants:
6. If of childbearing potential (WOCBP), the participant must agree, from Study Day 1 through 1 week after the last dose of study drug, to practice the protocol specified contraception. All WOCBP must have negative result of a serum pregnancy test performed at screening.

   a. Females of non-childbearing potential include postmenopausal (defined as age ≥ 55 years with no menses for 12 or more months without an alternative medical cause) or permanently sterile (e.g. bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
7. Participant voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB)-approved informed consent prior to performing any of the Screening Visit procedures.
8. Participant must be able to understand the nature of the study and must have the opportunity to have any questions answered

Exclusion Criteria:

1. Current clinically significant sleep disorder other than OSA of a severity that would interfere with study participation or interpretability of data.
2. Clinically significant craniofacial malformation or grade ≥3 tonsillar hypertrophy.
3. Current clinically significant cardiac disease (e.g., rhythm disturbances, coronary artery disease or cardiac failure) or poorly controlled hypertension (>140/90mmHg).
4. Long QT syndrome or family history of long QT syndrome
5. Current clinically significant neurological disorder, including epilepsy/convulsions.
6. Other active major organ system disease including renal failure, lung disease, neuromuscular disease, or liver disease.
7. Schizophrenia, schizoaffective disorder or bipolar disorder according to Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) or International Classification of Disease tenth edition criteria.
8. Attempted suicide within 1 year prior to screening, or current suicidal ideation.
9. Clinically significant urinary retention, gastric retention or other severe decreased gastrointestinal motility condition.
10. Benign prostatic hypertrophy that is actively being treated with alpha-1 adrenergic antagonist
11. Severe or frequent gastroesophageal reflux or constipation
12. Medically unexplained positive screen for drugs of abuse (excluding THC/marijuana) or history of substance use disorder as defined in DSM-V within 24 months prior to Screening Visit.
13. A serious illness or infection in the past 30 days as determined by investigator.
14. Clinically significant cognitive dysfunction as determined by investigator.
15. Untreated narrow angle glaucoma.
16. Women who are pregnant or nursing.
17. CPAP should not be used for at least 2 weeks prior to first study PSG and during entire participation in the study.
18. History of using oral or nasal devices for the treatment of OSA may enroll as long as the devices are not used for at least 2 weeks prior to first study PSG and during participation in the study.
19. History of using devices to affect participant sleeping position for the treatment of OSA, e.g. to discourage supine sleeping position, may enroll as long as the devices are not used for at least 2 weeks prior to first study PSG and during participation in the study.
20. Chronic oxygen therapy.
21. Patients with hypoglossal nerve stimulation implant. Prior/Concurrent Clinical Study Experience
22. Use of another investigational agent within 30 days or 5 half-lives, whichever is longer, prior to dosing.
23. Prolonged QT interval (> 450 ms in men or > 470 ms in women, after correction with most appropriate formula for observed heart rate), hypokalemia or hypomagnesemia (defined as >0.1 mEq/L below lower limit of normal for the testing laboratory).
24. Hepatic transaminases >2X the upper limit of normal (ULN), total bilirubin >1.5X ULN (unless confirmed Gilbert syndrome), estimated glomerular filtration rate < 50 ml/min.
25. Night- or shift-work sleep schedule which causes the major sleep period to be during the day, or planned travel across more than 1 time zone during the anticipated enrollment period
26. Employment as a commercial driver or operator of hazardous equipment.
27. Typically smoking more than 10 cigarettes or 2 cigars per day (or equivalent Vaping), or inability to abstain from smoking during overnight PSG visits.
28. Unwilling to use specified contraception.
29. History of regular alcohol consumption of more than 14 standard units per week (males) or more than 7 standard units per week (females), or unwillingness to limit alcohol consumption to no greater than 2 units/day (males), 1 unit per day (females). Alcohol is not to be consumed within 3 hours of bedtime or on PSG nights.
30. Unwilling to agree to limit during the study period caffeinated beverage intake (e.g., coffee, cola, tea) to 200 mg/day or less of caffeine, not to be used within 3 hours of bedtime. Viloxazine may increase the duration of effect of caffeine.
31. Any condition that in the investigator's opinion would present an unreasonable risk to the participant, or which would interfere with their participation in the study or confound study interpretation.
32. Participant considered by the investigator, for any reason, an unsuitable candidate to receive viloxazine or AD816 components, or unable or unlikely to understand or comply with the dosing schedule or study evaluations.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopnea index (AHI) 4%, AD816 vs. Placebo | 14 days of treatment dosing per crossover arm (collected at the end of treatment dosing per crossover arm)
  Apnea-hypopnea index based on 4% hypopnea desaturation

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Farkas, MD, Study Director — Apnimed Inc.
Locations (3):
- United States (3):
  - Santa Monica Clinical Trials, Los Angeles, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Clayton Sleep Institute, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aishah A, Kim M, Gell L, Vena D, Azarbarzin A, Pho H, Norman D, Ojile J, Esmaeili N, Taranto-Montemurro L, Wellman A, Sands S, Messineo L. Effect of viloxazine and trazodone in obstructive sleep apnoea: a randomised, placebo-controlled, cross-over study. Thorax. 2025 Aug 15;80(9):641-649. doi: 10.1136/thorax-2024-222513. PMID 40360261